CLINICAL TRIAL: NCT05971459
Title: A Study of the Efficacy of IAMT as an Assessment Tool for Prediction of Progression of Parkinson's Disease
Acronym: Music Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wilfrid Laurier University (Other)
Responsible Party: Principal Investigator, Demian Kogutek, Assistant Professor, Wilfrid Laurier University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10013143
Record Dates: First submitted 2023-07-11; First posted 2023-08-02 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
Keywords: music therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Mixed-method group comparative study, individuals with PD vs healthy individuals
Who Masked: Participant
Masking Description: Participants will receive a standardized functional and cognitive evaluation, as well as gait, fine motor, and gross motor assessments. Functional status will be measured using the Short Physical Performance Battery and the Timed Up & Go Test (TUG) for basic and instrumental activities of daily living. Global cognition will be assessed using the Mini Mental State Examination (MMSE), the Montreal Cognitive Assessment (MoCA), the Trail-Making Test (TMT) A & B, the WAIS-R Digit Symbol Substitution Test (DSST), the Digit Span Test, and the Letter Number Sequencing test. Fine and gross motor skills will be assessed using the Action Research Arm Test, the Hydraulic Hand Dynamometer Test, the Box and Block Test (BBT), and the 9-Hole Pegboard Test (9HPT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individuals with PD (Experimental): One music therapy session of 30 minutes
  Interventions: Behavioral: Improvised Active Music Therapy
- Healthy Individuals (Active Comparator): One music therapy session of 30 minutes
  Interventions: Behavioral: Improvised Active Music Therapy

INTERVENTIONS:
Behavioral: Improvised Active Music Therapy — During the music improvisation process, the accredited music therapist will carefully listen to the participant's initial musical expression, including tempo, rhythmic structure, dynamics, and beat. The accredited music therapist will then join, reflecting or confirming aspects of the participant's musical expression using standard music therapy improvisation techniques such as mirroring, matching, dialoguing, and containing on their electronic instrument. By comparing the participant's and therapist's musical responses over the sessions, it will be possible to identify note frequency, velocity of movement, synchronization, and acquisition of rhythmic complexity.

SUMMARY:
The primary objective of this proposal is to examine the efficacy of Improvised Active Music Therapy (IAMT) sessions as an early novel tool for cognitive and motor assessment for individuals with Parkinson's Disease (PD) in neurological rehabilitation. This will be achieved by identifying subtle variations in how participants play music and correlating these data with mobility and cognitive parameters. The secondary objective is to examine and understand the participants' experience of playing improvised music through post-session interviews as a qualitative measure. We propose to conduct a mixed-method, single-blinded, age-matched group comparison of 25 older adults (= 50 years) with PD and 25 healthy older adults (= 50 years) at the Conrad Institute for Music Therapy Research (CIMTR), Faculty of Music, Wilfrid Laurier University. The CIMTR laboratory contains Musical Instrument Digital Interface (MIDI) equipment/instruments and MATLAB software, which will be used to collect and analyze the music data to compare the two groups. The long-term goal is to build a database of sessions to use Improvised Active Music Therapy (IAMT) as a complementary, reliable, and feasible assessment tool to predict whether older adults with PD will progress to Parkinson's Disease Dementia (PDD) or Dementia with Lewy Bodies (DLB) and distinguish the motor phenotype as Tremor Dominant (PDTD), Mixed (PDM), or Postural Instability and Gait Disturbances (PIGD).

The purpose of this project is to understand the effect of music therapy sessions on cognition and motor skills within the reciprocal improvised music interactions between music therapist and clients. Therefore, the specific objectives are as follows:

1. To examine how physical characteristics of different neurological conditions influence music measures (note frequency, velocity of movement, synchronization, and acquisition of rhythmic complexity).
2. To examine how music measures contribute to cognitive and motor performance.
3. To assess the contributions of individual difference factors such as diagnoses, hand dominance, musical training, music preference, participant's personal experience, and cognitive abilities to music involvement.

DETAILED DESCRIPTION:
All participants will be scheduled to come to the testing rooms at the Manfred and Penny Conrad Institute for Music Therapy Research (CIMTR) Improvisation Laboratory for participation. After the study is explained, questions are answered, and informed consent is obtained, the individual will complete the experiment.

At the beginning of the study, participants will receive a standardized functional and cognitive evaluation, as well as gait, fine motor, and gross motor assessments at the CIMTR lab. Additionally, a detailed demographic history will be taken, and prescription and over-the-counter medications will be recorded. Functional status will be measured using the Short Physical Performance Battery and the Timed Up & Go Test (TUG) for basic and instrumental activities of daily living. Global cognition will be assessed using the Mini Mental State Examination (MMSE), the Montreal Cognitive Assessment (MoCA), the Trail-Making Test (TMT) A & B, the WAIS-R Digit Symbol Substitution Test (DSST), the Digit Span Test, and the Letter Number Sequencing test. Fine and gross motor skills will be assessed using the Action Research Arm Test, the Hydraulic Hand Dynamometer Test, the Box and Block Test (BBT), and the 9-Hole Pegboard Test (9HPT).

Following the standardized functional and cognitive evaluation, gait, and fine and gross motor assessments, participants will undergo one individual IAMT assessment session consisting of 30 minutes of uninterrupted improvised music at the CIMTR. Participants will play music on a simplified electronic drum set (Roland TD-11K V-Compact Kit) with two drum pedals, two drum pads, and two cymbals. The supervised student or accredited music therapist will facilitate the session with an electric piano (Korg 88-Key) or guitar with MIDI outputs. MIDI files will be recorded with LogicPro (music software) and processed using MATLAB. The quantitative music outcomes provided by IAMT will allow us to objectively correlate them with functional and cognitive parameters.

During the music improvisation process, the supervised student or accredited music therapist will carefully listen to the participant's initial musical expression, including tempo, rhythmic structure, dynamics, and beat. The supervised student or accredited music therapist will then join, reflecting or confirming aspects of the participant's musical expression using standard music therapy improvisation techniques such as mirroring, matching, dialoguing, and containing on their electronic instrument. Mirroring involves playing exactly what the participant is playing. Matching is playing music that fits the participant's style. Dialogue is the process of free communication through musical play, allowing the therapist to introduce new musical material. Containing involves creating stable music that supports the participant's music. The supervised music therapy student or accredited music therapist will also incorporate call and response techniques and familiar music within the improvised music. At this stage, the primary goal will be to meet or blend with the participant's music. The supervised student or accredited music therapist will maintain these clinical improvisation techniques throughout the sessions. By comparing the participant's and therapist's musical responses over the sessions, it will be possible to identify note frequency, velocity of movement, synchronization, and acquisition of rhythmic complexity.

Following the music therapy session, the supervised student or accredited music therapist will conduct a post-session debrief of approximately 15 minutes. This will involve open-ended and closed-ended questions related to how participants felt during the music therapy session, their thoughts during the session, and their thoughts about the music played by the supervised music therapy student or accredited music therapist, as well as their own music playing.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 50 years old, of any gender and location, and have a clinical diagnosis of Parkinson's Disease (PD).
* Participants should be able to understand and communicate in English.
* Participants should be capable of walking independently for a distance of 80 meters, with or without the use of a gait aid (e.g., walker, cane).
* Participants should be able to sit independently for 30 minutes at a time.
* Participants should be willing to play on a drum-set.
* Participants should NOT be deemed cognitively impaired, as indicated by a score of greater than 24 out of 30 on the Montreal Cognitive Assessment (MOCA).

Exclusion Criteria:

* Individuals who are unable to understand or communicate in English.
* Individuals with any other neurological disorder that has residual motor deficits (e.g., epilepsy, multiple sclerosis).
* Individuals who are using psychotropic medications that can affect motor performance (e.g., neuroleptics/anti-psychotics, anti-convulsants, and benzodiazepines).
* Individuals who have experience as a musician or are currently learning to play an instrument.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Musical Interface Digital Instruments music measures | 30 minutes (same session) Note frequency + velocity = musical engagemnet measure
  Subtle variations in how participants play music: note frequency

SECONDARY OUTCOMES:
Musical Interface Digital Instruments music measures | 30 minutes (same session) Velocity + note frequency = musical engagemnet measure
  Subtle variations in how participants play music: velocity of movement

OTHER OUTCOMES:
Debriefing | 15 minutes
  Post-session interviews as a qualitative measure

CONTACTS AND LOCATIONS:
Locations (1):
- Wilfrid Laurier University, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
All data collected in the study will be retained for a period of 10 years after the completion of the study. After this time, the study data will be disposed of following the confidential shredding and recycling system implemented at Wilfrid Laurier University for the destruction of medical records.